CLINICAL TRIAL: NCT00558480
Title: A Double Blind, Placebo Controlled Randomized Trial of Vitamin A Supplementation for Modulation of Mycobacterium Tuberculosis Immune Responses in Children Aged 5-14 Years With Latent Tuberculosis.
Brief Title: Vitamin A Supplementation for Modulation of Mycobacterium Tuberculosis Immune Responses in Latent Tuberculosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council Unit, The Gambia (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Department of State for Health and Social Welfare, The Gambia (Other Government)
Responsible Party: Professor Tumani Corrah, Unit Director, MRC (UK) Laboratories
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: SCC 1066
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Latent Tuberculosis Infection
MeSH Terms: conditions — Latent Tuberculosis | interventions — Vitamin A; retinol palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Vitamin A
  Interventions: Drug: Vitamin A
- 2 (Placebo Comparator): Vitamin A placebo
  Interventions: Drug: Vitamin A placebo

INTERVENTIONS:
Drug: Vitamin A — Vitamin A capsules, as retinol palmitate 200,000 IU at enrollment, 3 and 6 months
  Other Names: Retinol Palmitate
  Arms: 1
Drug: Vitamin A placebo — Vitamin A placebo at enrollment, 3 and 6 months
  Arms: 2

SUMMARY:
In populations with high prevalence of latent tuberculosis infection (LTBI), malnutrition (PEM) may influence incident rates of TB. PEM and specific micronutrient deficiencies compromise cell mediated immunity (CMI) and increase susceptibility to, or severity of infections. Vitamin A supplementation significantly reduces all-cause child mortality. The mechanism of the benefits of supplementation on clinical outcomes is largely unknown, but is likely to be related to an influence on the immune system. Vitamin A supplementation promotes lymphogenesis and induces a higher proportion of CD4 naïve T-cells in children. Most cases of LTBI that progress to active disease are vitamin A deficient. Vitamin A deficiency is common in most TB endemic countries. At the MRC, 32% of TBCC contacts were vitamin A deficient.

Hypothesis:

The investigators plan to test the hypotheses: that supplementation with vitamin A will affect the magnitude and quality of immune responses to mycobacterial antigens and progression to clinical disease.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a significant global health problem. Approximately a third of the world's populations are infected with Mycobacterium tuberculosis and 95% of cases occur in developing countries. This enormous pool of latently infected individuals is expected to pose a major obstacle for TB control in highly endemic countries and globally. In high income, low TB burden countries, targeted testing of TB case contacts and treatment for latent TB infection (LTBI) is practised as a component of TB control strategies. However, this is not practised in high burden, low-income countries. New evidence from mathematical modelling suggests that, to meet millennium development goals, interventions against M. tuberculosis infection will be required.

Children are at increased risk of rapid progression to active disease (usually within a year for infants). , Malnutrition has been identified as a major risk factor for progression to TB because of its profound effect on cellular immune function- the key host defence against TB. There are 2 types of risk associated with malnutrition: acquisition of infection and risk of infection progressing to disease. Therefore, in populations with high prevalence of latent TB infection, co-prevalent malnutrition may influence TB incidence rates.

Vitamin A supplementation has been clearly shown to reduce all-cause child mortality in developing countries. Vitamin A given at recommended doses has a profound effect on improving outcomes in measles and overall childhood mortality and morbidity. The mechanism for this has been attributed to its modulation of immune responses in addition to correcting underlying deficiency.

In TB patients, it is nearly impossible to determine nutritional status before disease and thus determine whether malnutrition led to TB or TB led to malnutrition. However, some studies have established a link between vitamin A deficiency and susceptibility to respiratory infections and progression from latent to active TB disease. Preschool children with symptomatic vitamin A deficiency have been found to have respiratory disease at twice the rate in non-deficient children, irrespective of anthropometric status. Getz et al found 81% of persons in a cohort with LTBI that had low levels of vitamin A developed disease compared to 30% of those with normal levels. We had previously observed a 32% prevalence of vitamin A deficiency in a subset of Tuberculosis case contact study contacts with latent TB (unpublished data). The mechanism of the benefits of vitamin A on clinical outcomes especially as related to measles is largely unknown and on tuberculosis is yet to be proven. However, it is likely to be related to an influence on the immune system.In experimental and animal models, vitamin A promotes differentiation and cytokine secretion by macrophages and may down regulate the secretion of pro-inflammatory cytokines e.g. TNF-alpha and IL-6. in children. Vitamin A supplementation has been reported to promote lymphogenesis and induce a higher proportion of CD4 naïve T-cells (CD4+ CD45RA). In addition, the quality of T-cell function may also be affected by Vitamin A.There are data indicating that IFN-gamma production is decreased in vitamin A deficient children while optimal in normal children. Immune responses of PBMCs from non-deficient children stimulated with specific antigens were biased towards more of IFN-gamma, and less of IL-10 and IL-4. This cytokine profile is reminiscent of decreased Treg differentiation and/or Th1-type immune response induced by vitamin A, which is required for protection against an intracellular pathogen such as M.tb. Indeed, data from our previous studies suggest that initial decrease in Treg induction in contacts of TB cases was associated with protection against progression to TB disease

To the best of our knowledge we are unaware of any trial of vitamin A for modulation of immune responses associated with progression to active disease in children with latent TB. We will conduct a parallel group comparison of a dose of 200,000 IU Vitamin A supplementation or placebo in latently infected children aged 5-14 years to evaluate qualitative and quantitative modulation of T-cell responses and clinical disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy children aged 5-14 years
* Resident in the Greater Banjul area
* Normal chest X-ray
* Mantoux result ≥ 10mm in the widest diameter
* Positive T-SPOT-TB
* Negative HIV antibody test
* Negative pregnancy test for 12-14 year-old females

Exclusion Criteria:

* History of previous TB or treatment for TB
* Clinical case TB
* Current participation in another clinical trial (except SCC 1041, 1034)
* Clinically significant history or evidence of skin disorders, allergy, immunodeficiency, organ-specific disorders causing immunodeficiency.
* Likelihood of travel away from the study area during or for the duration of the study.
* Chronic use (≥14 days) of any oral or systemic steroid or use of other immunosuppressive/ immunomodulating agents.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of cytokine (IFN-gamma, IL-10, TNF-alpha, TGF-beta) levels produced in response to M. tb. | 2 years

SECONDARY OUTCOMES:
FoxP3 gene expression with RT-PCR on mRNA from PBMCs. | 2 years
Incidence of probable/confirmed TB; change in weight (mean weight gain) | 2 years
Qualitative (positive/negative) and quantitative (mean change in counts) reversion of the T-cell assay | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ifedayo MO Adetifa, MD FWACP, Principal Investigator — MRC (UK) Laboratories, The Gambia; Martin OC Ota, MD FWACP PhD, Principal Investigator — MRC (UK) Laboratories, The Gambia

REFERENCES:
- See also: Related Info — http://www.mrc.gm